CLINICAL TRIAL: NCT06616922
Title: Assessment of the Effects and Tolerability of RD03/2016 (Levofloxacin; Ketorolac Trometamol 0.5+0.5% w/v Eye Drops Solution) for the Treatment of Bacterial Conjunctivitis in Adults: a Multicentre, Randomized, Blinded-assessor, Phase II Non Inferiority Study - MIRAKLE
Brief Title: Assessment of the Effects and Tolerability of RD03/2016 for the Treatment of Bacterial Conjunctivitis in Adults
Acronym: MIRAKLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEVOKETO_02-2020
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Conjunctivitis, Bacterial
Keywords: RD03/2016; Levofloxacin
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Levofloxacin; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, blinded-assessor study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test arm (Experimental): Patients will be randomly assigned (1:1) to one of the two treatment groups
  Interventions: Drug: RD03/2016 eye drops
- Standard drug arm (Active Comparator): Patients will be randomly assigned (1:1) to one of the two treatment groups
  Interventions: Drug: Levofloxacin 0.5% eye drops solution (Oftaquix®)

INTERVENTIONS:
Drug: RD03/2016 eye drops — 1 drop, 4 times a day (approximately every 4 hours while awake) for 5 days starting from Day 1.
  Other Names: Levofloxacin + Ketorolac Trometamol 0.5+0.5% w/v eye drops solution
  Arms: Test arm
Drug: Levofloxacin 0.5% eye drops solution (Oftaquix®) — 1 drop, 8 times a day (approximately every 2 hours while awake) on Days 1 and 2, and 1 drop, 4 times a day (approximately every 4 hours while awake) on Days 3 through 5.
  Other Names: Oftaquix® 5 mg/ml eye drops solution
  Arms: Standard drug arm

SUMMARY:
This is a phase II, randomized, parallel-group, blinded-assessor, multicentre study to assess the non-inferiority of RD03/2016 eye drops vs. levofloxacin eye drops alone (1:1) in microbiological eradication in patients with a clinical diagnosis of bacterial conjunctivitis with moderate/severe signs.

DETAILED DESCRIPTION:
This study will enroll 252 patients with clinical diagnosis of acute bacterial conjunctivitis with moderate/severe signs (score ≥ 2 for each cardinal sign, i.e., bulbar conjunctival injection, palpebral conjunctival injection and conjunctival discharge).

Enrolled patients will attend three study visits: baseline (Day 0), On-Therapy (OT; Day 3-4) and final visit (Day 7-9). The duration of the study for each patient will be 7-9 days.

Enrolled patients will undergo the following assessments: anamnesis; ophthalmological examination; swab of the lower conjunctiva for bacteriological examination, and a urine pregnancy test (for women of childbearing potential). Patients will be provided with a study smartphone to take photographs of the affected eye at home. Photographs will be taken by the person (a relative or a caregiver) assisting the patient and uploaded on the server of the study eCRF through eyePRO.net.

Test product (i.e. RD03/2016 - Levofloxacin; Ketorolac Trometamol 0.5+0.5% w/v eye drops solution) is the first fixed dose association between a quinolone antibiotic (i.e. levofloxacin) highly effective on the pathogenic bacteria that most frequently cause eye infections, and a nonsteroidal anti-inflammatory drug (NSAID) (i.e. ketorolac) highly effective in the control of signs and symptoms associated with inflammation.

The dosage proposed for RD03/2016 is one drop 4 times a day for 5 days, lower than that currently approved for levofloxacin alone. In patients with clinical diagnosis of bacterial conjunctivitis and in presence of moderate/severe signs and symptoms requiring an anti-inflammatory treatment for rapid symptomatic improvement, the use of RD03/2016 compared to treatment with levofloxacin alone could lead to a substantial simplification of the therapeutic regimen, without changing the rate of microbiological eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of patient to consent and provide signed written informed consent
2. Male or female aged ≥ 18 year.
3. Clinical diagnosis of acute bacterial conjunctivitis with moderate/severe signs (score ≥ 2 for each cardinal signs, i.e. bulbar conjunctival injection, palpebral conjunctival injection and conjunctival discharge, in at least one eye), not previously treated with antibiotics, steroids and nonsteroidal anti-inflammatory drugs (NSAIDs).
4. Able and willing to follow study procedures.
5. Availability of a person (a relative or a caregiver) to be trained for the execution of the photographic documentation required by the study and for the use of eyePRO.net.
6. Willing to interrupt the use of contact lenses for the entire duration of the study.

Exclusion Criteria:

1. Any acute ocular clinical disease other than bacterial conjunctivitis.
2. Any ocular surgery (including laser treatment) in the study eye within 30 days prior to study entry.
3. Any ocular (in the study eye) or systemic antimicrobial agents administered concurrently or within 3 days prior to study entry.
4. Any ocular (in the study eye) or systemic steroids or NSAIDs administered concurrently.
5. Pathological conditions or treatments that in the opinion of the Investigator may interfere with the efficacy and/or safety evaluations of the study (e.g. chronic blepharitis, glaucoma, moderate-severe dry eye).
6. Participation in previous clinical studies if less than 5 half-lives of the Investigational Medicinal Product (IMP) used have passed.
7. Hypersensitivity to the products, other quinolones, acetylsalicylic acid and other NSAIDs (due to potential for cross-sensitivity), or their excipients.
8. Contraindications to ocular treatment with levofloxacin and/or ketorolac.
9. Pregnancy or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test at baseline visit and practice effective contraceptive measures throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with microbiological eradication | At the Final visit (Day 7-9)
  Absence/no growth of pathogenic microorganisms or reduction below pathogenic criteria of opportunistic microorganisms susceptible to levofloxacin identified at baseline, as assessed through bacteriological culture and antibiotic susceptibility testing at the final visit (Day 7-9).

SECONDARY OUTCOMES:
By-pathogen microbiological eradication rate of levofloxacin-susceptible bacteria | At baseline that are eradicated at the final visit (Day 7-9)
  Proportion of levofloxacin-susceptible pathogenic bacteria at baseline that are eradicated at the final visit (Day 7-9).
Overall per-patient microbiological eradication rate of bacteria intermediate or resistant to levofloxacin | At the final visit (Day 7-9)
  Proportion of patients (pooling both treatment groups) with microbiological eradication (i.e., absence/no growth of pathogenic microorganisms or reduction below pathogenic criteria of opportunistic microorganisms) of bacteria intermediate or resistant to levofloxacin at baseline (as assessed through bacteriological culture and antibiotic susceptibility testing), at the final visit (Day 7-9).
Overall by-pathogen microbiological eradication rate of bacteria intermediate or resistant to levofloxacin | At baseline that are eradicated at the final visit (Day 7-9)
  Proportion of pathogenic bacteria intermediate or resistant to levofloxacin at baseline (pooling both treatment groups) that are eradicated at the final visit (Day 7-9).
Proportion of patients with clinical cure | At Day 3-4 and final visit (Day 7-9)
  Absence or at least one-unit improvement vs. baseline of all cardinal signs of bacterial conjunctivitis (conjunctival discharge, bulbar conjunctival injection and palpebral conjunctival injection) at OT visit (Day 3-4) and final visit (Day 7-9).
Time to clinical cure | Every 12 ± 1 hours from Day 0 to Day 7-9
  Absence or at least one-unit improvement vs. baseline of all cardinal signs of bacterial conjunctivitis (conjunctival discharge, bulbar conjunctival injection and palpebral conjunctival injection), assessed through photographs taken every 12 ± 1 hours from Day 0 to Day 7-9, using the study smartphone and eyePRO.net.
Time to resolution (absence) of bacterial conjunctivitis symptoms | Every 12 ± 1 hours from Day 0 to Day 7-9
  Time to resolution (absence) of bacterial conjunctivitis symptoms (i.e. pain, burning/stinging, itching, tearing, foreign body sensation, photophobia and discomfort) recorded by the patient every 12 ± 1 hours from Day 0 to Day 7-9 through the electronic patient diary.

OTHER OUTCOMES:
Safety: Adverse events throughout the study | Throughout the study, from Day 0 to Day 7-9
  The number of patients with adverse events, and the number and types of events will be recorded throughout the study
Local tolerability: Ocular itching/burning or discomfort related to study drug instillation | Twice a day, from Day 0 to Day 5
  Ocular itching/burning or discomfort related to study drug instillation, assessed by a Numeric Rating Scale (NRS) (0 = no itching/burning or discomfort to 10 = unbearable itching/burning or discomfort), through the electronic patient diary.
Compliance: Assessment of the number of instillations | From Day 1 to Day 5
  Number of study drug instillations, assessed through the electronic patient diary from Day 1 to Day 5
Feasibility: Microbiological eligibility rate | At the Final visit (Day 7-9)
  The proportion of screened patients with positive culture for levofloxacin-sensitive bacteria.
Feasibility: Patient confidence in using the study smartphone and eyePRO.net | At the Final visit (Day 7-9)
  Taking photographs of the study eye, as well as in following the picture-capturing procedure as per Investigator's instructions.
  The confidence of the patient in using the study smartphone and eyePRO.net is assessed through a questionnaire on the final visit (Day 7-9) by means of NRSs of 'Ease of using the smartphone', 'Ease of use of eyePRO.net', and 'Ease of following the picture-capturing procedures' (range 0-10, where 0 indicates 'very difficult' and 10 indicates 'very easy').
Feasibility part 1: Assessment of the mean number of pictures uploaded at a time through eyePRO.net | At the Final visit (Day 7-9)
  Mean timing of picture upload for each patient deemed suitable for clinical evaluation by the central team of blinded assessors.
Feasibility part 2: Assessment of the mean number of pictures uploaded at a time through | At the Final visit (Day 7-9)
  Mean the percentage of timely picture uploads for each patient deemed suitable for clinical evaluation by the central team of blinded assessors.
Feasibility part 3: Assessment of the mean number of pictures uploaded at a time through | At the Final visit (Day 7-9)
  Mean the percentage of uploaded pictures for each patient deemed suitable for clinical evaluation by the central team of blinded assessors.
Feasibility: Accuracy of photographic assessments of clinical cure against the gold standard direct ocular examination | At the Final visit (Day 7-9)
  Sensitivity, specificity, positive predictive value and negative predictive value of photographic assessments of clinical cure against the gold standard direct ocular examination at both the on-therapy and final visits

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, Prof., Principal Investigator — Ospedale San Raffaele IRCCS S.r.l.
Locations (41):
- Städtisches Klinikum Karlsruhe Augenklinik, Karlsruhe, Germany
- Italy (27):
  - A.O.U. Policlinico Consorziale di Bari, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale della Versilia, Camaiore
  - Centro Polispecialistico Achille Sicari, Carrara
  - Presidio Ospedaliero G. Rodolico - A.O.U. "Policlinico - Vittorio Emanuele", Catania
  - ASST Franciacorta - Ospedale di Chiari, Chiari
  - Clinica Oftalmologica Ospedale SS Annunziata, Chieti
  - Clinica Oculistica Azienda Ospedaliero-Universitaria Careggi di Firenze, Florence
  - Clinica Oculistica Azienda Ospedaliero - Universitaria Policlinico "G. Martino", Messina
  - ASST Fatebenefratelli Sacco - Istituto Fatebenefratelli e Oftalmico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - ASST Santi Carlo e Paolo, Milan
  - Clinica Oculistica Ospedale San Giuseppe, Milan
  - Ospedale Maggiore Policlinico - U.O. Oculistica Fondazione IRCCS Ca' Granda, Milan
  - Oculistica Ospedale G. Fogliani, Milazzo
  - U.O.S.C. Oculistica Az. Osp. di Rilievo Nazionale A. Cardarelli, Napoli
  - A.O.U. Policlinico P. Giaccone, Palermo
  - ARNAS Civico Di Cristina Benfratelli, Palermo
  - Presidio Ospedaliero di Cisanello - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Fondazione Policlinico Universitario - IRCSS Agostino Gemelli, Roma
  - IRCCS Fondazione G.B. Bietti, Roma
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - S.S. Annunziata di Savigliano, Savigliano
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale di Treviso, AULSS2 Treviso, Treviso
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Russia (8):
  - Regional Budgetary Institution of Healthcare "Ivanovo Regional Clinical Hospital", Ivanovo
  - Federal State Autonomous Institution "S.N. Fedorov National Medical Research Center "MNTK "Eye Microsurgery" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Educational Institution of High Professional Education "Moscow State Medical Stomatology University named after A.I.Evdokimov", Moscow
  - State Budgetary Institution "National Medical Research Center for Eye Diseases named after Helmholts" of the Ministry of Healthcare of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution of the Omsk Region "Clinical Ophthalmological Hospital named after V.P. Vykhodtsev", Omsk
  - LLC Sphera-Med, Saint Petersburg
  - Private Institution of Healthcare "Clinical hospital "RR-Medicine" of the city of Saint-Petersburg", Saint Petersburg
  - State Budgetary Healthcare Institution of Yaroslavl Region "Clinical Hospital #2", Yaroslavl
- Spain (5):
  - Sección De Cornea, Hospital Universitario La Paz, Madrid
  - Ophthalmology Unit Empresa Pública Hospital Costa del Sol, Marbella
  - Hospital La Fe Avenida de Fernando Abril Martorell, Valencia
  - Servicio De Oftalmología Hospital Universitario Rio Hortega, Valladolid
  - Servicio Oftalmología (Unidad Córnea Y Superficie Ocular) - Hospital do Meixoeiro Camino De Meixoeiro, Vigo